CLINICAL TRIAL: NCT02281279
Title: A Phase I/II Trial of Romidepsin, Rituximab and Lenalidomide (R3) in Relapsed/Refractory B Cell Lymphomas Including Transformed Follicular Lymphoma
Brief Title: Rituximab, Romidepsin, and Lenalidomide in Treating Patients With Recurrent or Refractory B-cell Non-Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1288; NCI-2014-02186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RM-FOL-PI-0034; MC1288 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Lenalidomide; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (rituximab, romidepsin, lenalidomide) (Experimental): Patients receive rituximab IV over 90 minutes on day 1; romidepsin IV over 4 hours on either day 1, days 1 and 8, or days 1, 8, and 15; and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: lenalidomide; Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of romidepsin and lenalidomide when combined with rituximab and to see how well this combination works in treating patients with B-cell non-Hodgkin lymphoma that has returned (recurrent) or did not respond to treatment (refractory). Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Romidepsin and lenalidomide may stop the growth of cancer cells by blocking enzymes needed for cell growth. Giving rituximab together with romidepsin and lenalidomide may be a better treatment for B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of the combination of romidepsin, rituximab and lenalidomide in patients with relapsed/refractory B-cell non-Hodgkin lymphoma (NHL). (Phase I) II. To assess the overall response rate (ORR) of this combination in patients with transformed follicular lymphoma (FL). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the toxicity and safety of romidepsin in combination with lenalidomide and rituximab.

II. To assess complete response rate (CR), progression free survival (PFS), and overall survival (OS) of this combination in patients with transformed FL.

TERTIARY OBJECTIVES:

I. To assess the impact of B-cell leukemia/lymphoma 2 (BCL2) mutations on ORR among patients treated with this combination.

II. To assess the impact of BCL2 mutations on PFS among patients treated with this combination.

OUTLINE: This is a phase I, dose-escalation study of romidepsin and lenalidomide followed by a phase II study.

Patients receive rituximab intravenously (IV) over 90 minutes on day 1; romidepsin IV over 4 hours on either day 1, days 1 and 8, or days 1, 8, and 15; and lenalidomide orally (PO) on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Histological confirmation of relapsed (recurrent after previous therapy[ies]) or refractory (no response to previous therapy[ies]) B-cell NHL; note: patients with small lymphocytic lymphoma (SLL) are eligible however patients with chronic lymphocytic leukemia (CLL) are not eligible
* PHASE II: Histological confirmation of transformation of FL lymphoma to diffuse large B cell lymphoma or aggressive lymphoma
* The biopsy confirming diagnosis can be up to 12 weeks prior to registration as long as there is no intervening therapy; note: if patient has had lymphoma treatment since previous biopsy, a biopsy should be repeated
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Measurable disease (at least 1 lesion of >= 1.5 cm in diameter) as detected by computed tomography (CT) or the CT images of the positron emission tomography (PET)/CT
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin =< ULN
* Alkaline phosphatase =< 3 x ULN unless due to direct lymphoma involvement, and then =< 5 x ULN
* Aspartate transaminase (AST) =< 3 x ULN unless due to direct lymphoma involvement, and then =< 5x ULN
* Calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula
* Magnesium >= 1.6 mg/dL
* Potassium >= 3.5 mg/dL
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS)® program
* Willing to be registered into the mandatory Revlimid REMS® program, and willing and able to comply with the requirements of the REMS® program
* If currently not on anticoagulation medication, willing and able to take aspirin (325 mg) daily; note: if aspirin is contraindicated, the patient may be considered for the study after if on therapeutic dose warfarin or low molecular weight heparin; patients unable to take any prophylaxis are not eligible
* Life expectancy >= 3 months
* Ability to complete medication diary by themselves or with assistance
* Ability to provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: during the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide tissue for central review and blood samples for correlative research purposes

Exclusion Criteria:

* Prior therapy with histone deacetylase (HDAC) inhibitors or immunomodulatory drugs (IMDs) (lenalidomide or thalidomide)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Active central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells that requires therapy
* Prolongation of corrected QT interval of > 480 ms
* Receiving any medications that prolong the corrected QT (QTc) and have a known risk for Torsades de pointes; note: providers should use caution with drugs with possible increased risk for Torsades de pointes; patient will be eligible if they can be taken off these medications prior to initiation of therapy and no less than 4 half-life of the medication
* Receiving any medications or substances that are strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5)
* Use of the following strong inhibitors are prohibited =< 7 days prior to registration

  * Boceprevir (Victrelis™)
  * Clarithromycin (Biaxin®, Biaxin XL®)
  * Conivaptan (Vaprisol®)
  * Grapefruit juice
  * Indinavir (Crixivan®)
  * Itraconazole (Sporanox®)
  * Ketoconazole (Nizoral®)
  * Lopinavir/ritonavir (Kaletra®)
  * Mibefradil
  * Nefazodone (Serzone®)
  * Nelfinavir (Viracept®)
  * Posaconazole (Noxafil®)
  * Ritonavir (Norvir®)
  * Saquinavir (Invirase®)
  * Telaprevir (Incivek®)
  * Telithromycin (Ketek®)
* Receiving any medications or substances that are inducers of CYP3A4
* Use of the following inducers are prohibited =< 12 days prior to registration

  * Avasimibe
  * Bosentan (Tracleer®)
  * Carbamazepine (Carbatrol®, Epitol®, Equetro™, Tegretol®, Tegretol-XR®)
  * Efavirenz (Sustiva®)
  * Modafinil (Provigil®)
  * Phenobarbital (Luminal®)
  * Phenytoin (Dilantin®, Phenytek®)
  * Rifabutin (Mycobutin®)
  * Rifampin (Rifadin®)
  * St. John's wort
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known positivity for human immunodeficiency virus (HIV); note: baseline testing for HIV is not required
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; note: patients with hepatitis B and C are eligible at the discretion of the treating physician; appropriate counseling regarding the risks of rituximab should be provided
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy requiring therapy; exceptions: non-melanotic skin cancer or any cancer that in the judgment of the investigator will not interfere with treatment plan and response assessment; patients with >= 25% of the bone marrow radiated for other diseases are not eligible
* History of myocardial infarction =< 6 months prior to registration, unstable angina, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* History of life threatening or recurrent thrombosis/embolism; patients may participate if they are on anticoagulation during the treatment
* Receiving erythroid stimulating agents (erythropoietin [EPO]: Procrit, Aranesp)
* History of allogeneic bone marrow or stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
MTD, defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) (Phase I) | 28 days
Overall response rate (Phase II) | Up to 5 years
  A success is defined as a CR or partial response (PR) noted as the objective status. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Adverse events profile, graded according to the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | Up to 30 days post-treatment
  The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Toxicity profile, defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment (Phase I) | Up to 30 days post-treatment
  Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Response profile, defined to be a CR or PR noted as the objective status (Phase I) | Up to 5 years
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population.
CR rate (Phase II) | Up to 5 years
  Will be estimated by the number of patients who achieve a CR divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true complete response rate will be calculated.
Survival time (Phase II) | Time from registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
PFS (Phase II) | Time from registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
  The distribution of PFS will be estimated using the method of Kaplan-Meier.
Incidence of adverse events, graded according to the revised NCI CTCAE version 4.0 (Phase II) | Up to 30 days post-treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
BCL-2 sequence | Baseline
  Will be assessed as mutation present vs. absent. The correlation between overall response (responder vs. non-responder) and mutation status will be evaluated using Fisher's exact test. The PFS in each group will be estimated using the Kaplan-Meier method. The differences in PFS between the two mutation groups will be assessed using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Nowakowski, Principal Investigator — Mayo Clinic